CLINICAL TRIAL: NCT02545504
Title: A Phase 3 Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of GS-5745 Combined With mFOLFOX6 as First Line Treatment in Patients With Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Brief Title: Andecaliximab With mFOLFOX6 as First Line Treatment for Advanced Gastric or Gastroesophageal Junction Adenocarcinoma
Acronym: GAMMA-1
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GS-US-296-1080; 2015-001526-42 (EudraCT Number)
Record Dates: First submitted 2015-09-08; First posted 2015-09-10 (Estimated); Results first posted 2020-04-28 (Actual); Last update posted 2020-05-26 (Actual); Status verified 2020-05

CONDITIONS: Gastric Adenocarcinoma
Keywords: Gastroesophageal junction (GEJ); Stomach cancer
MeSH Terms: conditions — Stomach Neoplasms | interventions — andecaliximab; Leucovorin; Fluorouracil; Oxaliplatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Andecaliximab (Experimental): Andecaliximab plus mFOLFOX6 (LV+5-FU+OXA) during Cycles 1-6, followed by andecaliximab plus LV+5-FU during subsequent cycles
  Interventions: Drug: Andecaliximab; Drug: Leucovorin; Drug: 5-fluorouracil; Drug: Oxaliplatin
- Placebo (Placebo Comparator): Placebo plus mFOLFOX6 (LV+5-FU+OXA) during Cycles 1-6, followed by placebo plus LV+5-FU during subsequent cycles
  Interventions: Drug: Placebo; Drug: Leucovorin; Drug: 5-fluorouracil; Drug: Oxaliplatin

INTERVENTIONS:
Drug: Andecaliximab — 800 mg administered intravenously on Days 1 and 15 of each 28-day treatment cycle
  Other Names: GS-5745
  Arms: Andecaliximab
Drug: Placebo — Administered intravenously on Days 1 and 15 of each treatment cycle
  Arms: Placebo
Drug: Leucovorin — Administered intravenously per standard of care on Days 1 and 15 of each treatment cycle
  Other Names: LV
Drug: 5-fluorouracil — Administered intravenously per standard of care on Days 1 and 15 of each treatment cycle
  Other Names: 5-FU
Drug: Oxaliplatin — Administered intravenously per standard of care on Days 1 and 15 of each treatment cycle
  Other Names: OXA

SUMMARY:
The primary objective of this study is to compare the efficacy of andecaliximab (GS-5745) versus placebo in combination with modified fluorouracil (5-FU), leucovorin (LV), and oxaliplatin (OXA) (mFOLFOX6) as measured by overall survival.

ELIGIBILITY:
Key Inclusion Criteria:

* Adults with histologically confirmed adenocarcinoma of the stomach or gastroesophageal junction that is inoperable, locally advanced or metastatic and not amenable to curative therapy
* Adequate hematologic, liver, coagulation and kidney function
* Eastern Cooperative Oncology Group (ECOG) ≤ 1
* Evaluable disease per Response Evaluation Criteria in Solid Tumors (RECIST) v 1.1

Key Exclusion Criteria:

* Previous chemotherapy for locally advanced or metastatic gastric cancer.
* Human Epidermal Growth Factor Receptor 2 (HER2)-positive gastric cancer
* HIV, hepatitis B virus (HBV), or hepatitis C virus (HCV) infection
* Pregnant or breast feeding women
* Individuals with known or suspected central nervous system metastases or individuals requiring chronic daily treatment with oral corticosteroids
* Grade ≥ 2 peripheral neuropathy

Note: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 432 (Actual)
Dates: Start 2015-10-13 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2019-05-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gilead Study Director, Study Director — Gilead Sciences
Locations (134):
- United States (31):
  - Scripps Green Hospital, La Jolla, California
  - University of Southern California, Los Angeles, California
  - UCLA Jonsson Comprehensive Cancer Center, Los Angeles, California
  - Innovative Clinical Research Institute, Whittier, California
  - Cancer Center of Central Connecticut, Plainville, Connecticut
  - Omega Research Consultants LLC, DeBary, Florida
  - Edward Hospital & Health Services, Naperville, Illinois
  - Parkview Hospital, Fort Wayne, Indiana
  - Indiana University Goshen Center for Cancer Care, Goshen, Indiana
  - Ochsner Clinic Foundation, New Orleans, Louisiana
  - New England Cancer Specialists, Scarborough, Maine
  - Karamanos Cancer Institute, Detroit, Michigan
  - HCA Healthcare, Kansas City, Missouri
  - Carol G. Simon Cancer Center, Morristown, New Jersey
  - Regional Cancer Care Associates LLC - Sparta, Sparta, New Jersey
  - Weill Cornell Medical College - New York Presbyterian Hospital, New York, New York
  - University of Rochester, Rochester, New York
  - Duke Cancer Institute, Durham, North Carolina
  - Oncology Hematology Care, Inc., Cincinnati, Ohio
  - The Ohio State Medical Center, Columbus, Ohio
  - Northwest Cancer Specialists, Portland, Oregon
  - Charleston Hematology Oncology Associates, Charleston, South Carolina
  - Prairie Lakes Health Care System INC, Watertown, South Dakota
  - Tennessee Oncology, Nashville, Tennessee
  - Center for Cancer Blood Disorders, Fort Worth, Texas
  - The University of Texas MD Anderson Cancer Center, Houston, Texas
  - Texas Oncology-Seton Williamson, Round Rock, Texas
  - Scott and White Memorial Hospital, Temple, Texas
  - Utah Cancer Specialists, Salt Lake City, Utah
  - Virginia Commonwealth University, Richmond, Virginia
  - Virginia Mason Seattle Main Clinic, Seattle, Washington
- Australia (10):
  - The Canberra Hospital, Garran, Australian Capital Territory
  - Chris O'Brien Lifehouse, Camperdown, New South Wales
  - The Crown Princess Mary Cancer Centre, Westmead, New South Wales
  - Princess Alexandra Hospital, Brisbane, Queensland
  - Ashford Cancer Centre, Kurralta Park, South Australia
  - Royal Hobart Hospital, Hobart, Tasmania
  - Epworth Healthcare, Richmond, Victoria
  - Western Health Sunshine Hospital, St Albans, Victoria
  - The Tweed Hospital, Tweed Heads
  - Sydney Adventist Hospital, Wahroonga
- Belgium (2):
  - Centre Hospitalizer De L'Ardenne, Libramont, Chevigny
  - University Hospital Gent Department of Gastroenterology, Ghent
- Chile (3):
  - Instituto Nacional Del Cancer, Santiago
  - Instituto Clinico Oncologico del Sur, Temuco
  - Hospital Clinico Vina Del Mar, Viña del Mar
- Colombia (4):
  - Oncomedica S.A, Montería, Departamento de Córdoba
  - Dundacion Oftalmologica de Santander Clinica Ardila Lulle La Foscal, Floridablanca
  - Hospital Pablo Tobon Uribe, Medellín
  - Centro Medico Imbanaco de Cali S.A, Valle
- Czechia (5):
  - Fakultni Nemocnice Brno, Brno
  - Fakultni nemocnice Hradec Kralove, Hradec Králové
  - University Hospital - Czech, Olomouc
  - Thomayer Hospital, Prague
  - Oblastni Nemocnice Pribram, Příbram
- France (6):
  - CHU Jean Minjoz, Besançon
  - CHRU de Brest, Hopital Morvan, Institut de Cancerologie et d'Hematologie, Brest
  - Hôpitaux Civils de Colmar, Colmar
  - Institut Paoli Calmettes, Marseille
  - CHU de Nice-l Archet, Nice
  - CH Annecy-Gennevois, Pringy
- Germany (10):
  - Klinikum rechts der Isar Technical University of Ismaninger, Munich, Bavaria
  - Kliniken Nordoberpfalz AG, Weiden, Bavaria
  - DRK Klinken Berlin Abteilungsleiter Chiurgische Okologie, Berlin
  - Universitätsklinikum Carl Gustav Carus, Dresden
  - Kliniken Essen Mitte Studiensekretariat Onkologie Evang. Huyssens-Stiftung, Essen
  - Krankenhaus Nordwest gGmbH Institut für Klinisch Onkologische Med Klinik II, Frankfurt
  - Cancer Center Heilbronn-Franken, SLK-Kliniken, Heilbronn
  - Zentrum fur Innere Medizin Stauferklinikum Schwab, Mutlangen
  - Staedtisches Klinikum Muenchen Bogenhausen, München
  - Universitatsklinikum Ulm, Ulm
- Hungary (6):
  - Egyesített Szent István és Szent László Kórház -Rendelőintézet, Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Human Klinikai Vizsgalatok Regisztracios Kozpont - HKVRK, Győr
  - Pandy Kalman Hospital, Gyula
  - Borsod County Hospital Clinical Oncological and Radiotheraputic Center, Miskolc
  - Zala Megyei Korhaz Pozva Diabetes Kulsokorhaz, Zalaegerszeg
- Italy (7):
  - University Hospital Company of Pisana, Pisa, PI
  - Ente Ospedaliero Ospedali Galliera, Genova
  - IRCCS A.O.U. San Martino, Genova
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Ospedale San Raffaele, Milan
  - S.C. Oncologia Medica Azienda Ospedaliera Valtellina e Valchiavenna Presidio Ospedaliero di Sondrio, Sondrio
  - Azienda Ospedaliera Treviglio Caravaggio U.O. Oncologia Medica, Treviglio
- Peru (3):
  - Centro de Investigacion Instituto de oncologia y Radiotherpia de la Clinica, San Isidro, Lima region
  - Centro Medico monte Carmelo, Arequipa
  - Clinica Anglo Americana Calle Alfredo Salazar, San Isidro
- Poland (7):
  - Beskidzkie Oncology Center, Bielsko-Biala
  - Wojewodzki Szpital Zespolony w Elblagu Oddzial Onkologiczny, Elblag
  - Wielkopolskie Centrum Onkologii, Poznan
  - Mrukmed Lekarz Beata Madej Mruk i Partner Spolka Partnerska Oddzial Nr 1 w Rzeszowie, Rzeszów
  - Wojewodzki Szpital Zespolony im L Rydygiera w Toruniu, Torun
  - Klinka Gastroenterologii Okologicznej Centrum Okologii Instytut, Warsaw
  - Wojskowy Instytut Medyczny, Warsaw
- Romania (7):
  - Medisprof srl Oncologie P TA, Cluj-Napoca, Judet Cluj
  - Fundeni Clinical Institute, Bucharest
  - GRAL Medical SRL, Bucharest
  - Centrul de Oncologie Sfantul Nectarie SRL, Oncologie, Craiova
  - Sc Oncolab Srl, Craiova
  - SC Centrul de Oncologie Euroclinic SRL, Oncologie, Iași
  - Spitalul Judetean De Urgenta Sf Ion Cel Nou Suceava Sectia Oncologie Medicala Bdul, Suceava
- Spain (14):
  - Hospital Universitario de A Coruna C, A Coruña
  - Hospital Clinic de Barcelona, Barcelona
  - Hospital Del Mar Servicio de Oncologia, Barcelona
  - Hospital Parc Tauli, Barcelona
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Institut Catala de la Salut, Barcelona
  - Hospital General Universitario Gregorio Maranon, Madrid
  - Hospital Ramon y Cajal, Madrid
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Puerta de Hierro, Madrid
  - Hospital Regional Universitario de Malaga, Málaga
  - Hospital Universitario Morales Meseguer, Murcia
  - Complejo Hospitalario de Navarra, Pamplona
  - Hospital Virgen de Valme, Seville
- Turkey (Türkiye) (14):
  - Cukurova Universitesi, Adana
  - Ankara University Medical Faculty Ibni Sina Hospital, Ankara
  - Hacettepe Universitesi Tip Facultesi Cocuk Saligi ve Hastaklikleri Anabilim Dali, Ankara
  - Hacettepe University, Ankara
  - University of Uludag, Bursa
  - Trakya University, Edirne
  - Bezmialem University Hospital, Istanbul
  - Bezmialem Vakif Universitesi Tip Fakultesi Hastanesi, Istanbul
  - Istanbul Universitesi Onkoloji Enstitusu Medikal Onkoloji Bilim Dali, Istanbul
  - Marmara University, Kadıköy
  - Izmir Universitesi Hastanesi Yeni Girne Vulvari, Karşıyaka
  - Kocaeli Universty, Kocaeli
  - Inonu Universitesi Turgut Ozal Tip Merkezi Elazi, Malatya
  - Van Yuzuncu Yil Universitesi Tip Kaultesi Ic Hastaliklari Anabilim Dali Tibbi Okoloji Bilim Dali, Van
- United Kingdom (5):
  - New Queen Elizabeth Hospital, Birmingham
  - Peterborough City Hospital Peterborough and Stamford Hospitals NHS Foundation Trust, Cambridge
  - Royal Marsden Hospital Mulberry House, London
  - University College London, London
  - Christie Hospital NHS Foundation Trust, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Shah MA, Bodoky G, Starodub A, Cunningham D, Yip D, Wainberg ZA, Bendell J, Thai D, He J, Bhargava P, Ajani JA. Phase III Study to Evaluate Efficacy and Safety of Andecaliximab With mFOLFOX6 as First-Line Treatment in Patients With Advanced Gastric or GEJ Adenocarcinoma (GAMMA-1). J Clin Oncol. 2021 Mar 20;39(9):990-1000. doi: 10.1200/JCO.20.02755. Epub 2021 Feb 12. PMID 33577358

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at study sites in Australia, Europe, Chile, Colombia, Peru, Turkey, and the United States. The first participant was screened on 13 October 2015. The last study visit occurred on 15 May 2019.
Pre-assignment Details: 635 participants were screened.
Groups:
- Andecaliximab + mFOLFOX6: Participants were randomized to receive andecaliximab 800 mg intravenous (IV) plus mFOLFOX6 [leucovorin (LV)+5-fluorouracil (5-FU) + oxaliplatin (OXA)] IV as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by andecaliximab 800 mg IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 161.7 weeks.
- Placebo + mFOLFOX6: Participants were randomized to receive placebo IV plus mFOLFOX6 (LV+5-FU+OXA) as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by placebo IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 112.3 weeks.
Period: Overall Study
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Started | 218 | 214
Completed | 0 | 0
Not Completed | 218 | 214
Not completed — Death | 174 | 168
Not completed — Unknown reason | 30 | 32
Not completed — Withdrew consent | 9 | 11
Not completed — Investigator's discretion | 3 | 1
Not completed — Lost to Follow-up | 2 | 2

BASELINE CHARACTERISTICS:
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants.
Groups:
- Andecaliximab + mFOLFOX6: Participants were randomized to receive andecaliximab 800 mg IV plus mFOLFOX6 (LV+5-FU+OXA) IV as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by andecaliximab 800 mg IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 161.7 weeks.
- Total: Total of all reporting groups
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6 | Total
Number analyzed (Participants) | 218 | 214 | 432
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (11.9) | 61 (11.4) | 60 (11.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 61 | 111
  Male | 168 | 153 | 321
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Race: American Indian or Alaska Native | 0 | 1 | 1
    Race: Asian | 5 | 5 | 10
    Race: Black or African American | 4 | 4 | 8
    Race: White | 186 | 184 | 370
    Race: Not Permitted | 8 | 6 | 14
    Race: Other | 15 | 14 | 29
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Not Permitted = local regulators did not allow collection of race or ethnicity information.
  Participants
    Ethnicity: Hispanic or Latino | 38 | 32 | 70
    Ethnicity: Not Hispanic or Latino | 170 | 173 | 343
    Ethnicity: Not Permitted | 10 | 9 | 19
Region of Enrollment [Count of Participants; unit: Participants]
  Colombia | 5 | 6 | 11
  Romania | 15 | 13 | 28
  Hungary | 11 | 15 | 26
  United States | 47 | 59 | 106
  Czechia | 10 | 5 | 15
  United Kingdom | 5 | 6 | 11
  Spain | 27 | 28 | 55
  Turkey | 17 | 18 | 35
  Belgium | 2 | 3 | 5
  Poland | 13 | 11 | 24
  Italy | 8 | 6 | 14
  Australia | 13 | 18 | 31
  Chile | 15 | 11 | 26
  France | 10 | 3 | 13
  Peru | 4 | 4 | 8
  Germany | 16 | 8 | 24
Type of Cancer [Count of Participants; unit: Participants]
  Gastric | 142 | 143 | 285
  Gastroesophageal junction | 76 | 71 | 147

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival (OS)
Description: OS was defined as the time interval from the date of randomization to death from any cause.
Time Frame: Andecaliximab + mFOLFOX6 median follow-up at the time of final analysis: 19.43 months; Placebo + mFOLFOX6 median follow-up at the time of the final analysis: 19.45 months
Population: The Intent-to-Treat (ITT) Analysis Set included all randomized participants.
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Andecaliximab + mFOLFOX6: Participants were randomized to receive andecaliximab 800 mg IV plus mFOLFOX6 (LV+5-FU+OXA) IV as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by andecaliximab 800 mg IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 135.4 weeks at the time of final analysis.
- Placebo + mFOLFOX6: Participants were randomized to receive placebo IV plus mFOLFOX6 (LV+5-FU+OXA) as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by placebo IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 99.7 weeks at the time of final analysis.
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 218 | 214
months | 12.52 [11.2 to 14.0] | 11.76 [10.3 to 13.5]
Statistical Analysis 1: Comparison: Andecaliximab + mFOLFOX6 vs Placebo + mFOLFOX6; The primary and secondary endpoints were tested sequentially in the following gate-keeping order: the primary OS endpoint, then the secondary PFS endpoint, and finally the secondary ORR endpoint; Test type: Superiority; p = 0.5625, Log Rank — The significance level at final analysis is 0.046 (two-sided). Stratum with < 6 participants or no informative event by combined treatment arms was pooled with the smallest adjacent stratum for stratified analyses; p-value was stratified by Eastern Cooperative Oncology Group (ECOG) status, geographic region and primary tumor site; Cox Proportional Hazard = 0.93, 95% CI 2-sided [0.74 to 1.18] — Hazard ratio (HR) was stratified by ECOG status, geographic region and primary tumor site with treatment arm as the only covariate

2. Secondary Outcome: Progression-free Survival (PFS)
Description: PFS was defined as the interval of time from the date of randomization to the earlier of the first documentation of definitive disease progression or death from any cause.
Time Frame: Andecaliximab + mFOLFOX6 median follow-up at the time of the final analysis: 18.64 months; Placebo + mFOLFOX6 median follow-up at the time of the final analysis: 18.74 months
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 218 | 214
months | 7.46 [7.29 to 8.41] | 7.06 [5.52 to 7.46]
Statistical Analysis 1: Comparison: Andecaliximab + mFOLFOX6 vs Placebo + mFOLFOX6; The primary and secondary endpoints were tested sequentially in the following gate-keeping order: the primary OS endpoint, then the secondary PFS endpoint, and finally the secondary ORR endpoint. PFS was tested only if OS was significant. The P-value is for display only; Test type: Superiority; p = 0.1031, Log Rank — The significance level at final analysis was 0.032 (two-sided). Stratum with < 6 participants or no informative event by combined treatment arms was pooled with the smallest adjacent stratum for stratified analyses; p-value was stratified by ECOG status,geographic region and primary tumor site; Cox Proportional Hazard = 0.84, 95% CI 2-sided [0.67 to 1.04] — HR was stratified by ECOG status,geographic region;primary tumor site with treatment arm as a covariate.Stratum with <6 participants or no informative event by combined treatment arms was pooled with smallest adjacent stratum for stratified analyses

3. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was defined as the percentage of participants who achieve a complete response (CR) or partial response (PR) as assessed by Response Evaluation Criteria In Solid Tumors (RECIST) v1.1. CR was defined as the disappearance of all target lesions and disappearance of all non-target lesions and normalization of tumor marker level. PR was defined as at least a 30% decrease in the sum of diameters of target lesions, taking as reference the baseline sum diameters.
Time Frame: Up to 135.4 weeks at the time of final analysis
Population: Participants in the ITT Analysis Set were analyzed.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Andecaliximab + mFOLFOX6: Participants were randomized to receive andecaliximab 800 mg IV plus mFOLFOX6 (LV+5-FU+OXA) IV as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by andecaliximab 800 mg IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 135.4 weeks at the time of the final analysis.
- Placebo + mFOLFOX6: Participants were randomized to receive placebo IV plus mFOLFOX6 (LV+5-FU+OXA) as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by placebo IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 99.7 weeks at the time of the final analysis.
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 218 | 214
percentage of participants | 50.5 [43.6 to 57.3] | 41.1 [34.5 to 48.0]
Statistical Analysis 1: Comparison: Andecaliximab + mFOLFOX6 vs Placebo + mFOLFOX6; The primary and secondary endpoints were tested sequentially in the following gate-keeping order: the primary OS endpoint, then the secondary PFS endpoint, and finally the secondary ORR endpoint. ORR was tested only if OS and PFS were significant.The P-value is for display only; Test type: Superiority; p = 0.0493, Cochran-Mantel-Haenszel — [p-value comment as in outcome 2, analysis 1]; p-value was stratified by ECOG status, geographic region and primary tumor site; Odds Ratio (OR) = 1.47, 95% CI 2-sided [1.00 to 2.15] — OR was stratified by ECOG status, geographic region and primary tumor site. Stratum with < 6 participants or no informative event by combined treatment arms was pooled with the smallest adjacent stratum for stratified analyses
Statistical Analysis 2: Comparison: Andecaliximab + mFOLFOX6 vs Placebo + mFOLFOX6; The primary and secondary endpoints were tested sequentially in the following gate-keeping order: the primary OS endpoint, then the secondary PFS endpoint, and finally the secondary ORR endpoint. ORR was tested only if OS and PFS were significant; Test type: Superiority; ORR Difference = 9.4, 95% CI 2-sided [0.1 to 18.8] — The 2-sided 95% confidence interval (CI) of difference for ORR between the treatment and placebo is calculated based on stratum-adjusted Cochran-Mantel-Haenszel proportion

4. Secondary Outcome: Percentage of Participants Experiencing Treatment-emergent Adverse Events (TEAEs)
Description: An adverse event (AE) is any untoward medical occurrence in a clinical study participant administered a medicinal product, which does not necessarily have a causal relationship with the treatment. TEAEs are events in a given study period that meet any of the following criteria: Any AE with onset date of on or after andecalizimab/placebo start date and no later than 30 days after permanent discontinuation of all study treatment (andecaliximab/placebo and chemotherapy) or Any AEs with onset date of on or after the andecaliximab/placebo start date and no later than 55 days after permanent discontinuation of andecaliximab/placebo or AEs leading to discontinuation of andecaliximab/placebo.
Time Frame: First dose date up to the last dose date (maximum:161.7 weeks) plus 30 to 55 days
Population: The Safety Analysis Set included all participants who received at least one dose of andecaliximab/placebo.
Measure: Number; unit: percentage of participants
Groups:
- Andecaliximab + mFOLFOX6: Participants received andecaliximab 800 mg IV plus mFOLFOX6 (LV+5-FU+OXA) IV as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by andecaliximab 800 mg IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 161.7 weeks.
- Placebo + mFOLFOX6: Participants received placebo IV plus mFOLFOX6 (LV+5-FU+OXA) as per standard of care on Days 1 and 15 of each 28-day treatment cycle during Cycles 1-6, followed by placebo IV plus LV+5-FU on Days 1 and 15 during subsequent cycles until disease progression, unacceptable toxicity, consent withdrawal, or the participant's refusal of treatment for up to 112.3 weeks.
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 216 | 210
percentage of participants | 99.1 | 99.5

5. Secondary Outcome: Percentage of Participants With Clinically Relevant Treatment-emergent Laboratory Abnormalities
Description: Treatment-emergent laboratory abnormalities were graded per Common Terminology Criteria for Adverse Events (CTCAE), Version 4.03 where 0=None, 1=Mild, 2=Moderate, 3=Severe, 4=Potentially Life Threatening. Treatment-emergent laboratory abnormalities are defined as values that increase at least 1 toxicity grade from baseline at any post-baseline time point, up to 30 days after the last dose of all study treatment, or 55 days after the last dose of andecaliximab/placebo for participants who permanently discontinued all study treatments. If the relevant baseline laboratory value is missing, then any abnormality of at least Grade 1 was considered treatment-emergent.
Time Frame: First dose date up to the last dose date (maximum: 161.7 weeks) plus 30 to 55 days
Population: Participants in the Safety Analysis Set were analyzed.
Measure: Number; unit: percentage of participants
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
Number analyzed (Participants) | 216 | 210
percentage of participants
  Hematology | 94.4 | 89.5
  Serum Chemistry | 91.7 | 92.9
  Coagulation | 7.4 | 3.3

ADVERSE EVENTS:
Time Frame: All-Cause Mortality: First dose date up to 42 months; Adverse Events: First dose date up to the last dose date (maximum: 161.7 weeks) plus 30 to 55 days
Description: All-Cause Mortality:The Intent-to-Treat Analysis Set included all randomized participants.Serious Adverse Events and Other Adverse Events: The Safety Analysis Set included all participants who received at least one dose of andecaliximab/placebo.
Arm/Group | Andecaliximab + mFOLFOX6 | Placebo + mFOLFOX6
All-Cause Mortality (participants affected / at risk) | 174/218 | 168/214
Serious Adverse Events (participants affected / at risk) | 103/216 | 108/210
Other Adverse Events (participants affected / at risk) | 209/216 | 203/210
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab + mFOLFOX6 (N=216) | Placebo + mFOLFOX6 (N=210)
Anaemia (Blood and lymphatic system disorders) | 3 | 2
Disseminated intravascular coagulation (Blood and lymphatic system disorders) | 1 | 0
Febrile bone marrow aplasia (Blood and lymphatic system disorders) | 0 | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 6 | 5
Neutropenia (Blood and lymphatic system disorders) | 4 | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 2 | 1
Acute myocardial infarction (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0
Cardiac arrest (Cardiac disorders) | 1 | 3
Cardio-respiratory arrest (Cardiac disorders) | 2 | 1
Cardiovascular disorder (Cardiac disorders) | 1 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0
Pericarditis (Cardiac disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 7 | 8
Abdominal pain lower (Gastrointestinal disorders) | 1 | 0
Abdominal pain upper (Gastrointestinal disorders) | 2 | 2
Colitis (Gastrointestinal disorders) | 2 | 0
Constipation (Gastrointestinal disorders) | 3 | 2
Diarrhoea (Gastrointestinal disorders) | 3 | 5
Duodenal ulcer perforation (Gastrointestinal disorders) | 1 | 0
Dysphagia (Gastrointestinal disorders) | 3 | 3
Gastric haemorrhage (Gastrointestinal disorders) | 1 | 2
Gastric perforation (Gastrointestinal disorders) | 0 | 1
Gastric stenosis (Gastrointestinal disorders) | 0 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 6 | 4
Gastrointestinal obstruction (Gastrointestinal disorders) | 1 | 0
Gastrointestinal perforation (Gastrointestinal disorders) | 1 | 0
Gastrointestinal toxicity (Gastrointestinal disorders) | 1 | 0
Haematemesis (Gastrointestinal disorders) | 1 | 0
Ileus (Gastrointestinal disorders) | 1 | 1
Impaired gastric emptying (Gastrointestinal disorders) | 1 | 0
Incarcerated inguinal hernia (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 1 | 4
Intestinal pseudo-obstruction (Gastrointestinal disorders) | 0 | 1
Large intestinal obstruction (Gastrointestinal disorders) | 1 | 0
Melaena (Gastrointestinal disorders) | 2 | 1
Nausea (Gastrointestinal disorders) | 4 | 4
Obstruction gastric (Gastrointestinal disorders) | 3 | 6
Oesophageal perforation (Gastrointestinal disorders) | 1 | 0
Oesophageal stenosis (Gastrointestinal disorders) | 0 | 1
Oesophagitis (Gastrointestinal disorders) | 1 | 1
Pancreatitis acute (Gastrointestinal disorders) | 2 | 0
Small intestinal obstruction (Gastrointestinal disorders) | 2 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 4
Vomiting (Gastrointestinal disorders) | 11 | 8
Chest pain (General disorders) | 1 | 2
Death (General disorders) | 4 | 1
Fatigue (General disorders) | 0 | 2
General physical health deterioration (General disorders) | 4 | 3
Inflammation (General disorders) | 1 | 0
Mucosal inflammation (General disorders) | 0 | 1
Non-cardiac chest pain (General disorders) | 1 | 0
Pain (General disorders) | 1 | 0
Pyrexia (General disorders) | 3 | 4
Acute on chronic liver failure (Hepatobiliary disorders) | 1 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0
Cholangitis acute (Hepatobiliary disorders) | 0 | 1
Cholecystitis (Hepatobiliary disorders) | 1 | 0
Cholecystitis acute (Hepatobiliary disorders) | 1 | 0
Hepatic failure (Hepatobiliary disorders) | 1 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Anaphylactic reaction (Immune system disorders) | 0 | 1
Drug hypersensitivity (Immune system disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Appendicitis (Infections and infestations) | 0 | 1
Cellulitis (Infections and infestations) | 1 | 0
Diarrhoea infectious (Infections and infestations) | 0 | 1
Diverticulitis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 2 | 1
Lower respiratory tract infection (Infections and infestations) | 1 | 0
Neutropenic sepsis (Infections and infestations) | 1 | 0
Oesophageal candidiasis (Infections and infestations) | 0 | 1
Pneumonia (Infections and infestations) | 7 | 5
Pneumonia necrotising (Infections and infestations) | 0 | 1
Postoperative wound infection (Infections and infestations) | 1 | 0
Pyelonephritis acute (Infections and infestations) | 0 | 1
Respiratory tract infection (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 2 | 4
Septic shock (Infections and infestations) | 0 | 2
Staphylococcal infection (Infections and infestations) | 0 | 1
Upper respiratory tract infection (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 4 | 1
Urosepsis (Infections and infestations) | 0 | 1
Vascular device infection (Infections and infestations) | 0 | 1
Viral infection (Infections and infestations) | 1 | 0
Accidental overdose (Injury, poisoning and procedural complications) | 0 | 1
Anastomotic ulcer (Injury, poisoning and procedural complications) | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 1
Fibula fracture (Injury, poisoning and procedural complications) | 1 | 0
Hip fracture (Injury, poisoning and procedural complications) | 1 | 1
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1
Meniscus injury (Injury, poisoning and procedural complications) | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 0 | 1
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0
Spinal fracture (Injury, poisoning and procedural complications) | 1 | 0
Subcutaneous haematoma (Injury, poisoning and procedural complications) | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1
Alanine aminotransferase increased (Investigations) | 1 | 0
Aspartate aminotransferase increased (Investigations) | 2 | 0
Blood bilirubin increased (Investigations) | 0 | 1
Body temperature increased (Investigations) | 0 | 1
Electrocardiogram QT prolonged (Investigations) | 1 | 0
General physical condition abnormal (Investigations) | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 1 | 0
Occult blood positive (Investigations) | 0 | 1
Transaminases increased (Investigations) | 1 | 0
Weight decreased (Investigations) | 1 | 0
White blood cell count decreased (Investigations) | 1 | 1
Cachexia (Metabolism and nutrition disorders) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 3 | 3
Failure to thrive (Metabolism and nutrition disorders) | 1 | 0
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypoglycaemia (Metabolism and nutrition disorders) | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 0
Back pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 1
Osteolysis (Musculoskeletal and connective tissue disorders) | 0 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1
Metastases to meninges (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Oesophageal carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Tumour necrosis (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Carotid arteriosclerosis (Nervous system disorders) | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 1
Hydrocephalus (Nervous system disorders) | 0 | 1
Hypoaesthesia (Nervous system disorders) | 0 | 1
Neurological decompensation (Nervous system disorders) | 0 | 1
Peripheral sensory neuropathy (Nervous system disorders) | 1 | 0
Seizure (Nervous system disorders) | 0 | 1
Syncope (Nervous system disorders) | 2 | 1
Transient ischaemic attack (Nervous system disorders) | 0 | 1
Vocal cord paralysis (Nervous system disorders) | 0 | 1
Device dislocation (Product Issues) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 2 | 2
Nephritis (Renal and urinary disorders) | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1
Renal failure (Renal and urinary disorders) | 0 | 1
Urine flow decreased (Renal and urinary disorders) | 0 | 1
Prostatitis (Reproductive system and breast disorders) | 0 | 1
Acute respiratory distress syndrome (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 8 | 13
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 1 | 0
Swelling face (Skin and subcutaneous tissue disorders) | 0 | 1
Arteriosclerosis (Vascular disorders) | 0 | 1
Deep vein thrombosis (Vascular disorders) | 3 | 0
Embolism (Vascular disorders) | 0 | 1
Peripheral venous disease (Vascular disorders) | 0 | 1
Poor venous access (Vascular disorders) | 3 | 0
Venous thrombosis (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Andecaliximab + mFOLFOX6 (N=216) | Placebo + mFOLFOX6 (N=210)
Anaemia (Blood and lymphatic system disorders) | 61 | 62
Neutropenia (Blood and lymphatic system disorders) | 76 | 73
Thrombocytopenia (Blood and lymphatic system disorders) | 38 | 32
Abdominal distension (Gastrointestinal disorders) | 14 | 14
Abdominal pain (Gastrointestinal disorders) | 41 | 37
Abdominal pain upper (Gastrointestinal disorders) | 19 | 26
Ascites (Gastrointestinal disorders) | 11 | 13
Constipation (Gastrointestinal disorders) | 61 | 61
Diarrhoea (Gastrointestinal disorders) | 87 | 88
Dry mouth (Gastrointestinal disorders) | 8 | 12
Dyspepsia (Gastrointestinal disorders) | 20 | 8
Dysphagia (Gastrointestinal disorders) | 21 | 19
Flatulence (Gastrointestinal disorders) | 11 | 10
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 9 | 14
Nausea (Gastrointestinal disorders) | 106 | 118
Stomatitis (Gastrointestinal disorders) | 24 | 21
Vomiting (Gastrointestinal disorders) | 63 | 62
Asthenia (General disorders) | 62 | 52
Chest pain (General disorders) | 7 | 11
Fatigue (General disorders) | 79 | 72
Mucosal inflammation (General disorders) | 25 | 26
Oedema peripheral (General disorders) | 18 | 20
Pyrexia (General disorders) | 25 | 18
Temperature intolerance (General disorders) | 12 | 12
Upper respiratory tract infection (Infections and infestations) | 16 | 8
Urinary tract infection (Infections and infestations) | 16 | 11
Alanine aminotransferase increased (Investigations) | 11 | 12
Aspartate aminotransferase increased (Investigations) | 13 | 11
Blood alkaline phosphatase increased (Investigations) | 15 | 9
Neutrophil count decreased (Investigations) | 30 | 25
Platelet count decreased (Investigations) | 19 | 17
Weight decreased (Investigations) | 29 | 23
Decreased appetite (Metabolism and nutrition disorders) | 63 | 72
Dehydration (Metabolism and nutrition disorders) | 16 | 16
Hyperglycaemia (Metabolism and nutrition disorders) | 13 | 6
Hypoalbuminaemia (Metabolism and nutrition disorders) | 12 | 8
Hypokalaemia (Metabolism and nutrition disorders) | 28 | 22
Arthralgia (Musculoskeletal and connective tissue disorders) | 14 | 10
Back pain (Musculoskeletal and connective tissue disorders) | 25 | 20
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 12 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 11 | 4
Dizziness (Nervous system disorders) | 19 | 26
Dysaesthesia (Nervous system disorders) | 15 | 12
Dysgeusia (Nervous system disorders) | 21 | 15
Headache (Nervous system disorders) | 18 | 15
Neuropathy peripheral (Nervous system disorders) | 28 | 21
Neurotoxicity (Nervous system disorders) | 10 | 11
Paraesthesia (Nervous system disorders) | 27 | 24
Peripheral sensory neuropathy (Nervous system disorders) | 73 | 72
Taste disorder (Nervous system disorders) | 7 | 11
Insomnia (Psychiatric disorders) | 27 | 22
Cough (Respiratory, thoracic and mediastinal disorders) | 25 | 23
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 20 | 22
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 16 | 19
Hiccups (Respiratory, thoracic and mediastinal disorders) | 11 | 9
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 10 | 12
Alopecia (Skin and subcutaneous tissue disorders) | 14 | 16
Rash (Skin and subcutaneous tissue disorders) | 13 | 11
Hypertension (Vascular disorders) | 9 | 11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After conclusion of the study and without prior written approval from Gilead, investigators in this study may communicate, orally present, or publish in scientific journals or other media only after the following conditions have been met:

* The results of the study in their entirety have been publicly disclosed by or with the consent of Gilead in an abstract, manuscript, or presentation form; or
* The study has been completed at all study sites for at least 2 years

DOCUMENTS (2):
  • Study Protocol (2017-03-06): https://cdn.clinicaltrials.gov/large-docs/04/NCT02545504/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-03): https://cdn.clinicaltrials.gov/large-docs/04/NCT02545504/SAP_001.pdf